CLINICAL TRIAL: NCT03625635
Title: Effect of a Clinical Nutrition Intervention Program on Body Composition, Metabolism and Antioxidant Activity Associated With Micronutrients in Breast Cancer Patients During Antineoplastic Treatment
Brief Title: Effect of a Clinical Nutrition Intervention Program in Breast Cancer Patients During Antineoplastic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Humberto Francisco Astiazaran Garcia, PhD (Other)
Responsible Party: Sponsor-Investigator, Humberto Francisco Astiazaran Garcia, PhD, Director Department of Nutrition, Centro de Investigación en Alimentación y Desarrollo A.C.
Organization: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CE/005/2015
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Breast Neoplasm; Breast Cancer
Keywords: primary noninvasive breast cancer; sarcopenic obesity prevention; individualized nutrition intervention; food-based intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Masking during data analysis. Technicians and investigators will not be aware of the participants personal data and particularities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition diagnosis and intervention (Experimental): At baseline and 6-mo after, a nutrition diagnosis will be done by measuring body composition components with DXA and basic anthropometric measurements. Based on the results, an individualized food-based intervention will be prescribed for each patient according to her diagnosis, food preferences, cultural and socioeconomic status. Follow-up will be every 2-weeks and a different diet menu will be provided in each session by a specialized dietitian, unto 6-mo are completed and initial measurements are repeated.
  Interventions: Other: Individualized food-based intervention

INTERVENTIONS:
Other: Individualized food-based intervention — Diet plans and recommendations will be based on the individual's nutritional status, symptoms and treatment side-effects, socioeconomic and cultural preferences; as well as the WCRF/AICR guidelines adapting 1.5g/kg/d of dietary protein and when required, a caloric restriction (500-1000 kcal/d). Garlic and cruciferous vegetables will be encouraged as well as 5-9 servings of fruits and vegetables a day. The program will be based on the macronutrient meal-equivalent menu method, and standard food servings will be based on the Mexican Food Equivalent System. Breast cancer patients follow-up will be every 2-weeks and a different diet menu will be provided in each session by a specialized dietitian, unto 6-mo are completed.

SUMMARY:
The aim of this study is to evaluate the effect of a 6-mo individualized and specialized food-based nutrition intervention program in breast cancer patients' body composition, metabolism and antioxidant activity associated with micronutrients, during antineoplastic treatment.

It is a quasi-experimental prospective follow-up study of women with primary diagnosis of invasive breast cancer in Sonora, Mexico. Conducted between September 2015 through July 2018. The Ethics and Research Committees of The Oncology State Centre and the Food and Development Research Centre, have approved the study's protocol and procedures. At baseline, all participants must sign an informed consent form and answer an oral interview, including self-reported questionnaires, for their nutrition record.

At the beginning and 6-mo after, participants will be weighed during the morning in a digital scale and height will be measured using a digital stadiometer. Body mass index (BMI) will be calculated and classified according to the World Health Organization criteria. Waist and hip circumferences will be measured with a metal tape, according to the protocol of the International Society for the Advancement of Kinanthropometry (ISAK), by a certified anthropometrist. Body composition components will be measured in a dual-energy x-ray absorptiometry (Hologic Corporation 4500 Waltham, MA) by total body, L1-L4, and femur neck scans. Blood samples will be drawn by a certified phlebotomist using sterile equipment and aseptic techniques.

Breast cancer patients' total energy expenditure will be estimated using an algorithm for Mexican population. Diet plans and recommendations will be based on the individual's nutritional status, dietary habits, symptoms and treatment side-effects, socioeconomic and cultural preferences; as well as the WCRF/AICR guidelines adapting 1.5g/kg/d of dietary protein to avoid sarcopenic obesity and considering a caloric restriction (500-1000 kcal/d), when required. The individualized nutrition intervention program will be based on the macronutrient meal-equivalent menu method, and standard food servings will be based on the Mexican Food Equivalent System. To guarantee that the obtained content for each macronutrient (g/day) meets the theoretical calculations, protein ±1g/d, total fat ±1g/d, carbohydrates ±2g/d and energy ±15 kcal/d variations will be accepted.

Breast cancer patients follow-up will be every 2-weeks and a different diet menu will be provided in each session by a specialized dietitian, unto 6-mo are completed, and initial measurements will be repeated. The differences in body composition determinants will be analyzed using paired Student's t-test analysis for each variable. A two-tailed P-value of 0.05 or less will be considered significant.

Retinol, tocopherol and carotenoids determination will be performed using HPLC. Serum will be thawed and retinol will be extracted using chloroform:methanol (3:1) and hexane, extracted layers will be combined and then evaporated to dryness under a soft stream of nitrogen. Samples will be re-suspended in ethanol before injecting onto the HPLC using a YMC C-30 column (30 cm length, 4.6 mm internal diameter, 3 µm particle size and 100 mm pore size). The HPLC system is an Agilent 1200 with UV-Vis and PDA detectors. Commercial standards and internal standards will be used to assess concentration and extraction efficiency, respectively. Additionally, the investigators will use a standard NIST serum (National Institute of Standards and Technology; Gaithersburg, Maryland USA). The cut-off point for vitamin A deficient status will be set at < 1.05 μmol /L.

The plasma antioxidant capacity will be determined by the trolox-equivalent antioxidant capacity test (TEAC) and oxygen radical absorbance capacity assay (ORAC). For both assays, results will be expressed as millimoles of Trolox equivalents per liter. The effect and their interaction on the response variables will be determined by ANOVA. Tukey's test will be used for the comparison of the means. Values of p<0.05 will be accepted as statistically significant.

Human inflammatory cytokines and chemokines will be analyzed by using a panel of 12 pro-inflammatory cytokines as a conventional ELISA protocol all at once under uniform conditions. The cytokines and chemokines represented by this array will be IL1A, IL1B, IL2, IL4, IL6, IL8, IL10, IL12, IL17A, IFNg, TNFa, and GM-CSF.

Plasma activities of both enzymes, glutathione peroxidase (GPx) and superoxide dismutase (SOD) will be determined in baseline samples and after 6-mo, by using an ELISA (enzyme-linked immunosorbent assay) based upon a sandwich assay principle and can be used to detect levels of SOD as low as 0.066 ng/mL and 1.56 ng/mL for GPx.

ELIGIBILITY:
Inclusion Criteria:

* nonmetastatic breast cancer patient
* before antineoplastic treatment initiation

Exclusion Criteria:

* bone fracture(s)
* disease(s) that could affect body composition (i.e. hypothyroidism)
* disease(s) that would require an additional dietary therapeutic approach or consideration (i.e. diabetes)
* dietary supplement consumption
* body dimensions surpassed the equipment's capacity

Elimination Criteria:

* newly diagnosed disease(s) that could affect body composition (i.e. hypothyroidism)
* newly diagnosed disease(s) that would require an additional dietary therapeutic approach or consideration (i.e. diabetes)
* dietary supplement consumption during the intervention
* patient's decision to refuse or stop antineoplastic treatment
* patient's decision to quit the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Total body weight | baseline and after the 6-mo food-based intervention
  change in body weight (kilograms)

SECONDARY OUTCOMES:
Body fat mass | baseline and after the 6-mo food-based intervention
  change in body fat mass (kilograms)
Body fat-free mass | baseline and after the 6-mo food-based intervention
  change in fat-free mass (kilograms)
Skeletal muscle mass | baseline and after the 6-mo food-based intervention
  change in skeletal muscle mass (kilograms)
Waist circumference | baseline and after the 6-mo food-based intervention
  change in waist circumference (centimeters)
Retinol | baseline and after the 6-mo food-based intervention
  change in retinol μmol /L
Trolox-equivalent antioxidant capacity test | baseline and after the 6-mo food-based intervention
  change in trolox equivalents per liter
Glutathione peroxidase (GPx) | baseline and after the 6-mo food-based intervention
  change in glutathione peroxidase concentration (ng/mL)
Superoxide dismutase (SOD) | baseline and after the 6-mo food-based intervention
  change in superoxide dismutase concentration (ng/mL)
Human inflammatory cytokines | baseline and after the 6-mo food-based intervention
  change in IL1A, IL1B, IL2, IL4, IL6, IL8, IL10, IL12, IL17A, IFNg, TNFa, and GM-CSF (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Humberto Astiazaran-Garcia, PhD, Study Director — Centro de Investigacion en Alimentacion y Desarrollo (CIAD)
Locations (1):
- Centro de Investigacion en Alimentacion y Desarollo (CIAD), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Limon-Miro AT, Valencia ME, Lopez-Teros V, Aleman-Mateo H, Mendez-Estrada RO, Pacheco-Moreno BI, Astiazaran-Garcia H. An individualized food-based nutrition intervention reduces visceral and total body fat while preserving skeletal muscle mass in breast cancer patients under antineoplastic treatment. Clin Nutr. 2021 Jun;40(6):4394-4403. doi: 10.1016/j.clnu.2021.01.006. Epub 2021 Jan 9. PMID 33485708